CLINICAL TRIAL: NCT01489930
Title: Effects of Resistance and Endurance Training on Synthesis of Individual Muscle Proteins in Young and Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, K. Sreekumaran Nair, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 07-007689
Record Dates: First submitted 2011-11-18; First posted 2011-12-12 (Estimated); Last update posted 2011-12-12 (Estimated); Status verified 2011-12

CONDITIONS: Sarcopenia
Keywords: Exercise; Aging; Sarcopenia; Mitochondria
MeSH Terms: conditions — Sarcopenia; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Endurance Exercise (Experimental): Participants will perform 8-weeks of moderate intensity endurance (cycling) exercise
  Interventions: Behavioral: Endurance exercise
- Resistance Exercise (Experimental): Participants will perform 8-weeks of whole-body resistance exercise training.
  Interventions: Behavioral: Resistance exercise
- Control / Combined Training (Experimental): Participants will perform 8-weeks of no exercise, followed by an additional 8-weeks of combined endurance plus resistance exercise training.
  Interventions: Behavioral: Control/Combined training

INTERVENTIONS:
Behavioral: Endurance exercise — Participants will perform 8-weeks of endurance exercise training. Participants will train 5 days per week for 60 min at 65% of VO2 peak.
  Arms: Endurance Exercise
Behavioral: Resistance exercise — Participants will perform 8-weeks of resistance exercise training. Participants will train 4 days per week for ~60 min. Two days will focus on lower body resistance training and two days will focus on upper body.
  Arms: Resistance Exercise
Behavioral: Control/Combined training — Participants will perform 8-weeks of no exercise (control), followed by 8-weeks of combined endurance and resistance training. Participants will endurance train 5 days per week for 30 min at 65% of VO2 peak and resistance train 4 days per week for 30 min.
  Arms: Control / Combined Training

SUMMARY:
Loss of skeletal muscle strength and skeletal muscle mass occurs with of aging. This are-related decline in skeletal muscle mass and skeletal muscle strength is a major underlying factor contributing to many of the metabolic disorders and frailty of the investigators rapidly expanding aging population. Endurance (aerobic) and resistance exercise training programs have been shown to effectively reverse the age-related decline in metabolic and contractile muscle functions. The investigators will measure synthesis rates of individual muscle proteins in 36 each of young (18-30 yrs) and 36 older (> 65 yrs) people to determine their response to 8 weeks each of endurance, resistance, combined endurance and resistance training, or placebo exercise training.

Hypotheses.

1. to measure fractional synthesis rates of multiple muscle proteins and identify those that are enhanced by an endurance exercise program
2. to determine whether changes in protein synthesis in response to endurance exercise programs are dependent on age
3. to measure fractional muscle synthesis rates of multiple muscle proteins and to identify those that are enhanced by a resistance exercise program
4. to determine whether changes in protein synthesis in response to resistance exercise programs are dependent on age

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* 18 to 30 or >65 years
* Males and Females

Exclusion Criteria:

* Regular Exercise Program
* Smoking
* Cardiometabolic Disease (diabetes, cardiovascular disease, thyroid disorders)
* Drugs known to impair metabolic function (beta blockers, steroids)
* Allergies to lidocaine
* Physical disability that precludes exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2008-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Skeletal Muscle Protein Synthesis | Measured at week 0 (baseline) and week 8
  The investigators will determine the change from baseline in skeletal muscle protein synthesis. Measurments will be performed at baseline and following 8 weeks of exercise training.

SECONDARY OUTCOMES:
Mitochondrial Function | Measured at week 0 (baseline) and week 8
  The investigators will determine the change from baseline in mitochondrial function. Measurments will be performed at baseline and following 8 weeks of exercise training.

CONTACTS AND LOCATIONS:
Overall Officials: K. Sreekumaran Nair, MD, PD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Irving BA, Lanza IR, Henderson GC, Rao RR, Spiegelman BM, Nair KS. Combined training enhances skeletal muscle mitochondrial oxidative capacity independent of age. J Clin Endocrinol Metab. 2015 Apr;100(4):1654-63. doi: 10.1210/jc.2014-3081. Epub 2015 Jan 19. PMID 25599385